CLINICAL TRIAL: NCT01919606
Title: Evaluation of the Safety and Efficacy of EXPAREL(R) (Bupivacaine Liposome Injectable Suspension) When Administered Into the Transversus Abdominis Plane (TAP) for Prolonged Postoperative Analgesia in Subjects Undergoing Open Total Abdominal Hysterectomy
Brief Title: EXPAREL Administered Into the TAP for Analgesia in Subjects Undergoing Open Total Abdominal Hysterectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA402S23B703
Record Dates: First submitted 2013-02-26; First posted 2013-08-09 (Estimated); Results first posted 2014-05-14 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Postoperative Pain
Keywords: hysterectomy; analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EXPAREL Group 1 (Experimental): EXPAREL 266 mg diluted with saline to a volume of 40 mL
  Interventions: Drug: EXPAREL
- EXPAREL Group 2 (Experimental): EXPAREL 266 mg diluted with saline to a volume of 60 mL
  Interventions: Drug: EXPAREL

INTERVENTIONS:
Drug: EXPAREL — Single-dose EXPAREL diluted with 20 mL or 40 mL saline to a volume of 40 mL or 60 mL, respectively.
  Other Names: Bupivacaine liposome injectable suspension

SUMMARY:
The primary objective of this study is to determine the optimal of two different volumes of EXPAREL 266 mg when administered via infiltration into the transversus abdominis plane (TAP) for prolonged postoperative analgesia in subjects undergoing open total abdominal hysterectomy.

DETAILED DESCRIPTION:
This is a prospective, open-label, non-randomized study with two treatment groups differing only in the volume of EXPAREL infiltrated into the TAP. All subjects will undergo an open total abdominal hysterectomy. The dose of EXPAREL for the TAPs will be the same for all 20 subjects, 133 mg on the right side of the abdomen and 133 mg on the left side of the abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Females, 18-75 years of age inclusive.
* American Society of Anesthesiologist (ASA) physical status 1-3.
* Undergoing open total abdominal hysterectomy (i.e., laparoscopic procedures are not sufficient) without any concurrent surgical procedure(s).
* Physically and mentally able to participate in the study and complete all study assessments.
* Able to give fully informed consent to participate in this study after demonstrating a good understanding of the risks and benefits of the TAP.

Exclusion Criteria:

* Demonstrated hypersensitivity or idiosyncratic reactions to amide-type local anesthetics.
* Any subject whose anatomy, or surgical procedure, in the opinion of the Investigator, might preclude the potential successful performance of a TAP.
* Any subject who in the opinion of the Investigator might be harmed or be a poor candidate for participation in the study.
* Any subject, who in the opinion of the Investigator, is on chronic pain medicine.
* Subjects who have received any investigational drug within 30 days prior to study drug administration, or planned administration of another investigational product or procedure during their participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dorian, MD, Principal Investigator — St. Barnabas Medical Center, Livingston, NJ 07039; Thad Denehy, MD, Principal Investigator — St. Barnabas Medical Center, Livingston, NJ 07039

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EXPAREL Group 1 | EXPAREL Group 2
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EXPAREL Group 1 | EXPAREL Group 2 | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (0) |  | 67 (0)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 1 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Duration of Analgesia
Time Frame: End of surgery to time of subject's first postsurgical opioid administration (through 72 hours)
Arm/Group | EXPAREL Group 1 | EXPAREL Group 2
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Incidence of Adverse Events
Time Frame: 10 days post surgery plus or minus 3 days
Measure: Number; unit: number of events
Arm/Group | EXPAREL Group 1 | EXPAREL Group 2
Number analyzed (Participants) | 1 | 0
number of events | 0 |

ADVERSE EVENTS:
Time Frame: 10 days post surgery plus or minus 3 days
Description: Normal systematic assessment for adverse events
Arm/Group | EXPAREL Group 1 | EXPAREL Group 2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No